CLINICAL TRIAL: NCT03258905
Title: Phone App for Grounding (De-escalation) of Substance-abusing Transition-age Youth
Brief Title: Phone App for Grounding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Treatment Innovations (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R44AA026746-02A1 (NIH); R44AA026746-02A1 (NIH)
Record Dates: First submitted 2017-08-16; First posted 2017-08-23 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Substance-Related Disorders
Keywords: transition-age youth; mobile app; grounding; Seeking Safety
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grounding enhanced app (Experimental): A mobile app that uses the Seeking Safety grounding chapter content, enhanced with features designed to create strong engagement and interactivity
  Interventions: Behavioral: Grounding enhanced app
- Grounding text-only app (Active Comparator): A mobile app that uses the Seeking Safety grounding chapter content in text format only
  Interventions: Behavioral: Grounding text-only app

INTERVENTIONS:
Behavioral: Grounding enhanced app — A mobile app that uses the Seeking Safety grounding chapter content, enhanced with features designed to create strong engagement and interactivity
  Arms: Grounding enhanced app
Behavioral: Grounding text-only app — A mobile app that uses the Seeking Safety grounding chapter content in text format only
  Arms: Grounding text-only app

SUMMARY:
The goal of this project is to continue to develop a smartphone application ("app") to help youth from ages 18-25 who have a substance abuse problem. The app will engage them in grounding, which is a sensory-based experience to help them feel calm by reducing intense negative feelings and impulses (such as the urge to use a substance or hurt themselves or others).

DETAILED DESCRIPTION:
Substance use disorder (SUD) is the second most common psychiatric diagnosis in the U.S. population. Transition-age youth (TAY) from ages 18-25 are especially vulnerable to substance use and SUD. This time period represents a distinct stage separate from adolescence and later adulthood. It includes tasks such as leaving home to enter college, the workforce, or the military; clarifying vocational goals; and attaining legal drinking age. This period is also prime for experimentation with substance use and associated risks such as driving under the influence, accidents, fighting and violence, HIV, and vulnerability to sexual assault. This project focused on a major strategy, grounding, to help TAY de-escalate (reduce) intense negative emotions and impulses. Grounding has long been used in psychiatric hospitals to provide a safe, quick, and powerful way to reduce any intense negative feeling such as impulses to hurt self or others, substance craving, anger, anxiety, etc. Described in detail in the book Seeking Safety (SS), grounding using three pathways to focus the mind (mental), body (physical), and heart (soothing). Grounding provides a way to regulate emotion, which is a major challenge for TAY, especially given their hormone changes and emotional intensity. Indeed substance use is often described as a short-term way to regulate emotion. Grounding is a key module of SS, a widely-implemented, evidence-based SUD treatment model. In phase 1 the investigator developed a beta version of a grounding app. The app promotes the use of grounding in any environment in which emotions and impulses need to be regulated. It capitalizes on TAYs' widespread use of mobile devices; and because grounding is a stand-alone skill and sensory-oriented, it lends itself wonderfully to an app approach. An iterative product development methodology was used based on end-user feedback and the impact of the app was studied in a pilot randomized controlled trial (RCT) with 24 TAY. Half received the app and the other half received grounding handouts. Results showed that the app was consistently more positively rated than the handouts and was associated with significantly more use of grounding and a higher score on a grounding knowledge test. All phase 1 benchmarks were met. In phase 2 the investigator proposes to scale up both the app and the evaluation of it. There are two specific aims: (1) To enhance the mobile grounding app by using exciting, innovative technology approaches as well as expanding the grounding content in amount and type. (2) To conduct an RCT with 68 TAY to evaluate the grounding app versus a control app. The control app would control for both the use of a mobile device and the grounding content. The primary outcome is based on power analysis from the phase 1 pilot; other outcomes and measures are also included. The RCT uses rigorous scientific methods in its design, measures, and statistics.

ELIGIBILITY:
Inclusion Criteria:

* outpatient
* meets criteria for substance use disorder per the treatment site
* has a smartphone (either Android or iOS)
* has not attended and is not currently attending Seeking Safety treatment

Exclusion Criteria:

* current uncontrolled psychotic or bipolar disorder
* currently criminal-justice involved such that we would need to report substance use or other possible criminal behavior (e.g., to a parole or probation officer)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Grounding Knowledge Test | 6 weeks

SECONDARY OUTCOMES:
Total time spent on the app | 6 weeks
BASIS-32 Impulsive and Addictive Behavior subscale | 6 weeks
Difficulties in Emotion Regulation Scale | 6 weeks

OTHER OUTCOMES:
Brief Addiction Monitor | 6 weeks
Coping Self-Efficacy Scale | 6 weeks
BASIS-32 total score | 6 weeks
Perceived Stress Scale | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Najavits, PhD, Principal Investigator — Treatment Innovations
Locations (1):
- Treatment Innovations, Newton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No